CLINICAL TRIAL: NCT02122861
Title: A Phase 1, Open-Label Clinical Trial Evaluating the Safety, Tolerability and Immunogenicity of Intradermally Administered ID-LV305 in Patients With Locally Advanced, Relapsed, or Metastatic Cancer Expressing NY-ESO-1
Brief Title: Phase 1 Study of Intradermal LV305 in Patients With Locally Advanced, Relapsed or Metastatic Cancer Expressing NY-ESO-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID-LV305-2013-001
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Melanoma - Currently Enrolling; Non-small Cell Lung Cancer - Enrollment Completed; Sarcoma - Enrollment Completed
Keywords: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ID-LV305 (Experimental): Dose escalation and expansion cohort including treatment of melanoma
  Interventions: Biological: ID-LV305

INTERVENTIONS:
Biological: ID-LV305 — pembrolizumab

SUMMARY:
This is a Phase 1 multi-center study to evaluate the clinical safety and immune response of ID-LV305 when injected intradermally in patients with advanced cancer. ID-LV305 is a novel immunotherapy agent designed to target dendritic cells and stimulate the body's immune system to fight the spread and growth of cancer for patients whose tumors express the NY-ESO-1 protein. Patients with melanoma, sarcoma, ovarian cancer, or small cell lung cancer that express NY-ESO-1 may be considered for the trial. Selected sites will be evaluating ID-LV305 with pembrolizumab for patients with melanoma who have inadequately responded to anti-PD-1 therapy.

DETAILED DESCRIPTION:
ID-LV305 is an agent designed to specifically target dendritic cells within the patient and induce them to stimulate and generate cytotoxic T cell responses against the NY-ESO-1 protein, a molecule which is often expressed in certain types of cancer cells. This is a first in human study of ID-LV305. The primary purpose of the study is to determine what dose ID-LV305 can be given safely to patients with advanced cancers that express NY-ESO-1 protein. ID-LV305 will be administered by intradermal injection every three weeks times four doses. The study will have two phases. In Part 1, Dose Escalation, which has been completed, three sequentially enrolled cohorts of patients were treated at one of four dose levels of ID-LV305 using a standard escalation design. Followed by Part 2 expansion where an additional 27 subjects were enrolled. In Part 2SA, Site-specific Amendment, patients with unresectable and/or metastatic melanoma with an inadequate response to anti-PD-1 MAb therapy, defined as SD or PD using RECIST criteria following at least 2 months of therapy. Patients with PD have a tumor measurement increase of <2-fold from the time of starting anti-PD-1 therapy, must not be symptomatic or have worsening of Eastern Cooperative Oncology Group (ECOG) performance status due to their disease progression, and cannot have new CNS lesion. Patients must also meet the lactic acid dehydrogenase (LDH), ECOG status, and no tumor size criteria are used in Part 2SA.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, relapsed, and/or metastatic cancer with low or minimal tumor burden which may or may not be measurable; no tumor size criteria are used.
* Tumor histology consistent with melanoma tumor specimen positive for NY-ESO-1 expression by IHC and/or RT-PCR.
* b. In Part 2SA, patients with an inadequate response to anti-PD-1 mAb therapy, defined as SD or PD using RECIST v1.1 criteria following at least 2 months of therapy. Patients with PD have a tumor measurement increase of < 2 fold from the time of starting anti-PD-1 therapy, must not have worsening of Eastern Cooperative Oncology Group (ECOG) performance status due to their disease progression, and cannot have new CNS lesion. Patients must also meet the lactic acid dehydrogenase (LDH) or ECOG status. No tumor size criteria are used in Part 2SA.
* ≥ 18 years of age.
* Life expectancy of ≥ 6 months per the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* ECG without evidence of clinically significant arrhythmia or ischemia.
* If female of childbearing potential (FCBP), willing to undergo pregnancy testing and agrees to use at least one highly effective or two effective contraceptive methods during the dosing period and for three months after last LV305 injection. If enrolled on the arm that includes pembrolizumab, agrees to use highly effective contraceptive methods during the dosing period and for 120 days after last injection of study drug.
* If male and sexually active with a FCBP, must agree to use highly effective contraception such as latex condom during the dosing period and for three months after last LV305 injection. If enrolled on the arm that includes pembrolizumab, agrees to use highly effective contraceptive methods during the dosing period and for 120 days after last injection of study drug.

Exclusion Criteria:

* Investigational therapy within 3 weeks prior to LV305 dosing.
* Prior administration of other NY-ESO-1-targeting immunotherapeutics.
* Significant immunosuppression from:

  1. Concurrent, recent (≤ 4 weeks ago) or anticipated treatment with systemic corticosteroids at any dose, or
  2. Other immunosuppressive medications such as methotrexate, cyclosporine, azathioprine (antihistamines, non-steroidal anti- inflammatory drugs and aspirin permitted) or conditions such as common variable hypogammaglobulinemia or exposures such as large field radiotherapy
* Cancer therapies, including chemotherapy, radiation, biologics or kinase inhibitors, G-CSF or GM-CSF within 3 weeks prior to the first scheduled LV305 dosing. For patients enrolled in Part 2, Site-specific Amendment, erythropoietin, G-CSF, and GM-CSF will be allowed and anti-PD-1 therapy may be given within 3 weeks if it follows their prior treatment schedule.
* Psychiatric, other medical illness or other condition that in the opinion of the PI prevents compliance with study procedures or ability to provide valid informed consent.
* Significant autoimmune disease with the exception of alopecia, vitiligo, hypothyroidism or other conditions that have never been clinically active or were transient and have completely resolved and require no ongoing therapy. For patients enrolled in Part 2SA who have the potential to receive pembrolizumab, active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, etc.) is not considered a form of systemic treatment.
* Myocardial infarction within 6 months of study initiation, active cardiac ischemia or New York Heart Association (NYHA) Grade III or IV heart failure.
* Inadequate organ function including:

  1. Marrow: Peripheral blood leukocyte count (WBC) < 3000/mm3, absolute neutrophils count ≤ 1500/mm3, platelets < 75000/mm3, or hemoglobin < 10 gm/dL.
  2. Hepatic: alanine aminotransferase (ALT), and aspartate aminotransferase (AST) > 2.5 x ULN, total serum bilirubin > 1.5 x ULN (patients with Gilbert's Disease may be included if their total bilirubin is ≤ 3.0 mg/dL).
  3. Renal: Creatinine > 1.5x ULN.
  4. Other: INR (prothrombin time ratio) or partial thromboplastin time (PTT) >1.5 x ULN.
* For patients enrolled in Part 2SA who are receiving anti-PD-1 mAb therapy, marrow and hepatic function as defined in criteria 8a and 8b may be up to CTCAE Grade 2 if first reviewed, found to be within acceptable safety parameters for treatment with pembrolizumab, and approved by the Sponsor Medical Monitor.
* History of other cancer within 3 years (except non-melanoma cutaneous malignancies and cervical carcinoma in situ). For patients enrolled in Part 2 of the Site-specific Amendment, history of other cancer within 1 year (except non-melanoma cutaneous malignancies and cervical carcinoma in situ. Concurrent active cancers are not allowed).
* Active tuberculosis or recent (< 2 week ago) clinically significant infection or evidence of active hepatitis B, hepatitis C or HIV infection.
* Brain metastases considered unstable as:

  1. Without confirmed stability over 60 days in patients previously treated with prior surgery or radiation; OR
  2. Associated with symptoms and/or findings; OR
  3. Requiring corticosteroids or anticonvulsants in the prior 60 days
  4. If enrolled in Part 2SA, new, growing, or previously untreated lesions since the start of anti-PD-1 therapy.
* Pregnant, planning to become pregnant, or nursing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 5 years after first study vaccine injection.
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability].

SECONDARY OUTCOMES:
Immunogenicity | Approximately 12 weeks
  Measure changes from baseline in anti-NY-ESO-1 serum antibodies and anti-LV antibodies and changes from baseline in peripheral blood of NY-ESO-1 specific CD4+, CD8+, Teff and Treg cells.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (7):
- United States (7):
  - San Francisco Oncology Associates, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Dana Farber Harvard Cancer Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Greenville Health System, Greenville, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington